CLINICAL TRIAL: NCT06274320
Title: Investigation of the Effect of a 2 Weeks Lipikar Urea 30% Application Preceding a Planned Topical 5-FU 4% Actinic Keratoses Treatment on Efficacy of 5-FU 4%
Brief Title: Effect of Lipikar Urea 30% Before Actinic Keratoses Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: LRP22002 LIPIKAR UREA 30%
Record Dates: First submitted 2024-02-16; First posted 2024-02-23 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Actinic Keratoses
Keywords: actinic keratoses; Lipikar Urea 30%; Olsen grade
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: holistic approach (Experimental): adult subjects having AK (grade I or II) lesions on the scalp and meeting specific inclusion/exclusion criteria including a Tolak® treatment planned before study start
  Interventions: Other: Group A: holistic approach
- Group B: Tolak® Standard of use (Active Comparator): adult subjects having AK (grade I or II) lesions on the scalp and meeting specific inclusion/exclusion criteria including a Tolak® treatment planned before study start
  Interventions: Other: Group B: Tolak® Standard of use

INTERVENTIONS:
Other: Group A: holistic approach — 2-week Lipikar Urea 30% application (once daily in the evening) + 4-week Tolak® treatment (once daily in the evening)
  Arms: Group A: holistic approach
Other: Group B: Tolak® Standard of use — 4-week Tolak® alone treatment (once daily in the evening)
  Arms: Group B: Tolak® Standard of use

SUMMARY:
This study is conducted in one center in Germany, in adult subjects having actinic keratoses (grade I or II) lesions on the scalp and meeting specific inclusion/exclusion criteria. The purpose of the study is to evaluate a holistic management (efficacy, tolerability and lesion cosmetic outcomes) of Tolak® treatment.

DETAILED DESCRIPTION:
Actinic keratoses (AK) are chronic skin changes usually induced by UV radiation. There are numerous options to treat AK. Some of the most used field-directed therapies include topical therapy with 5-fluorouracil (5-FU) cream and photodynamic therapy. However, the treatment with 5-FU is not without side effects (erythema, pruritus, itching/burning, etc.). Therefore, in daily clinical practice, cosmetic pre- and concomitant applications of cosmetics are often recommended to increase the efficacy as well as the tolerability of Tolak®.

The aim of this randomized, evaluator blinded, controlled parallel group study conducted in compliance with the 2013 version of the Declaration of Helsinki is to determine whether and how the application of cosmetics leads to an influence on the microbiome of AK.

Statistical method: The variables will be analyzed by using the Cochran-Mantel-Haenszel (CMH) statistic, after ridit transformation with the row mean difference statistics, testing the hypothesis of equality. Each test will be two-sided, at the 0.050 significance level.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of at least 4 non-hypertrophic, non-hyperkeratotic actinic keratosis of the the scalp
* planned treatment of actinic keratoses of the scalp with Tolak®
* Olsen grade I or II

Exclusion Criteria:

* known or documented intolerance to any of the ingredients of Tolak® or Lipikar Urea 30%
* treatment of actinic keratoses in the treatment area within the past 3 months (e.g. photodynamic therapy, topical 5-FU, diclofenac, imiquimod, cryotherapy etc.)
* suspected invasive squamous cell cancer in the treatment area
* chronic wounds, erosions, pre-existing inflamed or infected skin with disruption of the epidermal barrier in the treatment area current or within the last 8 weeks given systemic cancer medication or systemic treatment with 5-Fluorouracil

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in lesion response rate | from baseline to Day70
  It is defined as the number of completely responding lesions divided by the total number of treated lesions in each field. Complete lesion response is defined as complete disappearance of the lesion both by palpation and visual.

SECONDARY OUTCOMES:
Percentage change | from baseline to Day70
  The lesion complete response rate is defined as the percentage of pre-existing and treated lesions at Baseline that are assessed as clear (complete disappearance of the lesion, visually and by palpation).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dirschka, Principal Investigator — CentroDerm GmbH
Locations (1):
- CentroDerm GmbH, Wuppertal, Germany